CLINICAL TRIAL: NCT03681002
Title: Implementation of a Structured Lifestyle Program in a Primary Care Setting. Changes in Lifestyle and Effects on Cardiovascular Risk in Patients With High Cardiovascular Risk.
Brief Title: Implementation of a Structured Lifestyle Program in Primary Care. Changes in Lifestyle Habits and Cardiovascular Risk.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DNR 2014/ 497
Record Dates: First submitted 2018-09-18; First posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Cardiovascular Risk Factor; Lifestyle Risk Reduction; Primary Care
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- structured lifestyle program (Other): individual counseling focusing on Lifestyle habits
  Interventions: Behavioral: structured lifestyle program

INTERVENTIONS:
Behavioral: structured lifestyle program — Intensive Lifestyle counseling during one year

SUMMARY:
The aim of the present study is to describe and evaluate the effect of a structured lifestyle intervention program, focusing on lifestyle habits, in a primary care setting in patients with high cardiovascular risk. Furthermore, we want to explore the patient´s experience of lifestyle change and counseling after participation in the intervention program and to investigate the cost-effectiveness of the program.

DETAILED DESCRIPTION:
Intervention The intervention program comprises five individual visits to the same nurse, specialised in diabetes care and the metabolic syndrome every three month during one year. The nurse led a person centered dialog based on the answers from a questionnaire. At every visit, focus was primarily on lifestyle habits, using motivational interviewing to strengthen the patient's ability to modify one or more lifestyle habits. Dietary counselling was in accordance with the Swedish recommendation in nutrition. If the patient were in need of extended counseling regarding one or more lifestyle habits, he or she could be referred within the primary care unit to a specialist. During the 12-month period, all patients where offered to participate in evening group sessions at three different occasions. Topics were physical activity, fatty acids, healthy food, tobacco and alcohol, stress, sleep and methods of how to change behavior".

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with

* hypertension
* diabetes mellitus type 2
* impaired glucose tolerance

Exclusion Criteria:

* dementia
* severe psychiatric disease
* difficulties to understand Swedish

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | From baseline to 12 months
  Patients rating perceived physical activity on a scale 0-10 at baseline and at 12 months

SECONDARY OUTCOMES:
Framingham risk score | From baseline to 12 months
  The Framingham Risk Score is a gender-specific algorithm used to estimate the 10-year cardiovascular risk of an individual. Cardiovascular risk scoring systems give an estimate of the probability that a person will develop cardiovascular disease within a specified amount of time, in this case 10 years. Individuals with low risk have 10% or less CHD risk at 10 years, with intermediate risk 10-20%, and with high risk 20% or more.

CONTACTS AND LOCATIONS:
Overall Officials: Mattias K Damberg, Principal Investigator — Associate professor, Department of Public health and caring sciences; Family medicine and preventive medicin

IPD SHARING:
Plan to Share IPD: Undecided